CLINICAL TRIAL: NCT04283968
Title: Clinical Efficacy of Fecal Microbial Transplantation Treatment in Adults With Moderate-to-Severe Atopic Dermatitis
Brief Title: Efficacy of Fecal Microbial Transplantation Treatment in Adults With Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TLV 0452-17
Record Dates: First submitted 2020-02-19; First posted 2020-02-25 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The care providers, investigators, outcome assessor, and the participants do not know which of the transplantations is placebo and which is fecal microbial one during the first phase of the study. After the 4 transplantations the patients of the placebo group will have the possibility to enter an open label study in which they will receive 4 fecal transplantations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): All patients will receive 4 fecal microbial transplantations from healthy donors each 2 weeks apart
  Interventions: Biological: Fecal Microbial Transplantation
- Placebo followed by treatment arm (Placebo Comparator): All patients will receive 4 placebo fecal transplantations followed by 4 fecal microbial transplantations from healthy donors each 2 weeks apart
  Interventions: Biological: Fecal Microbial Transplantation; Biological: placebo fecal transplantation

INTERVENTIONS:
Biological: Fecal Microbial Transplantation — Fecal Microbial Transplantation in adults with Atopic Dermatitis
Biological: placebo fecal transplantation — placebo fecal transplantation
  Arms: Placebo followed by treatment arm

SUMMARY:
Prospective double-blinded placebo-controlled study, among adult patients suffering from moderate-to-severe atopic dermatitis (AD), insufficiently responsive to topical and systemic treatment. In the first group all patients will receive 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. In the second group all patients will receive 4 placebo transplantations each 2 weeks apart. Patients will be allowed to continue with their baseline medical topical treatment, including moisturizers and glucocorticoids, during the study period, but no new therapy should be commenced. The patients of the second group, who received the placebo treatment will have the possibility to enter an open label phase in which they will receive 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. The severity of AD and the fecal microbiome profile will be evaluated by the Scoring Atopic Dermatitis Score (SCORAD score), Investigator Global Assessment scale for Atopic Dermatitis (IGA) and the weekly use of topical corticosteroids, at the beginning of the study, before every FMT, and 1-6 months after the last FMT.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, placebo-controlled study aimed to assess the safety and clinical efficacy of FMT for the treatment of mild-moderate AD, and to assess the change in the fecal microbiota following FMT in the study population. The study will include 2 groups. In the first group all patients will receive 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. In the second group all patients will receive 4 placebo transplantations each 2 weeks apart. Patients will be allowed to continue with their baseline medical topical treatment, including moisturizers and glucocorticoids, during the study period, but no new therapy should be commenced. The patients of the second group, who received the placebo treatment, will have the possibility to enter an open label phase in which they will receive 4 fecal microbial transplantations (FMTs) from healthy donors each 2 weeks apart. The clinical activity of AD, adverse events and the fecal microbiome profile will be evaluated at the beginning of the study, before every FMT, and 1-6 months after the last FMT, using the SCORAD score, the IGA assessment scale, and the weekly use of topical corticosteroids.

During the study period, patients will be allowed to use only topical therapy including emollients and glucocorticoids or calcineurin inhibitors.

FMT preparation and delivery:

Volunteer donors will be healthy, non-pregnant adults aged 18 to 50 years, with a normal body mass index. They will be excluded for any significant medical history or for any use of antibiotics in the preceding 3 months. Candidates should be eligible according to the Israeli Ministry of Health guidelines which include a physical examination and laboratory screening tests including fecal enteric pathogens, serum antibodies to hepatitis A, B, and C; human immunodeficiency virus; HTLV, and Treponema pallidum as well as celiac, CBC (and additional tests that comply with the guidelines of the Israeli Ministry of Health). Stool will be delivered within minutes post defecation in a clean closed plastic container and will be processed at the Tel Aviv Medical Center stool bank facility to prepare capsulized FMT. Briefly, fecal material will be diluted with normal saline (600ml/100g of fecal material), filtered and concentrated the preparation in a centrifuge. The pellet will be suspended in sterile saline and glycerol (20%) that will be added as a bacterial cryoprotectant. This material will be then pipetted into acid-resistant capsules, which will be closed and then secondarily sealed with additional set of capsules. Capsules will be stored frozen at -80°C. Placebo capsules will have identical visually and contained diluted glycerol only.

Capsulized FMT procedure:

FMT will be administered two doses of 15 FMT capsules on two consecutive days (a total of 30 capsules), at the Bacteriotherapy clinic of the Tel Aviv medical center (TLVMC). On the day of administration, capsules frozen at -80°C will be taken out of the freezer and transported to the clinic on ice. Fifteen capsules will be handed individually to the patient and the patient will ingest the capsules immediately with some water. Patients will be asked to fast overnight prior to capsule intake.

Fecal microbial analysis:

In order to examine whether the clinical effect may be mediated by colonization of new bacterial strains, we developed a robust and sensitive method to calculate pairwise DNA sequence dissimilarity between bacterial strains of the same species across distinct metagenomics samples. Donor stool samples that will be used for FMT capsules and stool samples that will be collected from the patients during the study period will be sequenced into metagenomics reads. Reads that will be mapped will be piled up to obtain per-position variant information for every detected species. Difference in the variant of a particular species at a given position between two samples will be defined as having no intersection between the set of detected alleles in the two samples being compared. The estimated species DNA sequence dissimilarity for a pair of samples is then the number of different positions divided by the total number of positions being compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥18 years of age, with moderate-to-severe atopic dermatitis, as defined by a Scoring Atopic Dermatitis Score (SCORAD) score ≥25, with disease duration minimum of 3 years that was inadequately controlled by topical and systemic therapy

Exclusion Criteria:

1. Age under 18 years
2. Pregnancy
3. Another concomitant active dermatologic disease.
4. Receiving systemic therapy including phototherapy within 4 weeks before the beginning of the study.
5. receiving any antibiotic or probiotic treatment within 2 weeks before the beginning of the study or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the change in the severity of Atopic Dermatitis after treatment with Fecal Microbial Transplantation | 2 weeks after each FMT, and 8 weeks or more after the last FMT
  Overall mean change from baseline of the Scoring atopic dermatitis score (SCORAD), described and validated by the European Task Force on Atopic Dermatitis, used for the assessment of the severity of Atopic Dermatitis. The minimal SCORAD score, describing a situation without any signs of atopic dermatitis is 0, the disease is not visible, while the maximal score, describing the most severe presentation of atopic dermatitis, is 103.

SECONDARY OUTCOMES:
Association between the improvement in disease severity and the degree of bacterial strain transmission from donor to patient. | 2 weeks after each FMT, and 8 weeks or more after the last FMT
  Assessment of the relation between the microbiome of donors and patients by calculating DNA sequence dissimilarity between bacterial strains of the same species across donor stool samples that were used for FMT capsules and stool samples that were collected from the patients during the study period.

OTHER OUTCOMES:
Assessment of the change in the IgE level after treatment with Fecal microbial transplantation | 2 weeks after each FMT, and 8 weeks or more after the last FMT
  Assessment of the change in the IgE level after treatment with Fecal microbial transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Mashiah, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Nitsan Maharshak, Study Director — Tel-Aviv Sourasky Medical Center
Locations (2):
- Israel (2):
  - Department of Dermatology, Tel Aviv Sourasky medical center, Tel Aviv
  - Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes
After termination of the study protocol for all participants the data and stool and blood samples will be shared in order to perform fecal microbial analysis to examine whether the clinical effect may be mediated by colonization of new bacterial strains
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After termination of the study protocol for all participants the data and stool and blood samples will be shared
Access Criteria: All information will be given to the researcher that will perform the fecal microbial analysis